CLINICAL TRIAL: NCT01147055
Title: A Phase 1, Fixed Sequence, Cross-Over Study To Estimate The Effect Of Multiple Dose Rifampin On The Single Dose Pharmacokinetics Of Crizotinib (PF-02341066) In Healthy Volunteers
Brief Title: Estimation Of Effect Of Rifampin On Pharmacokinetics Of Crizotinib In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: A8081016
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2011-10-19 (Estimated); Last update posted 2011-10-24 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: crizotinib; healthy volunteers; rifampin; pharmacokinetics; single dose
MeSH Terms: interventions — Crizotinib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): There should be at least 14-day washout period between treatment A and B.
  Interventions: Drug: crizotinib; Drug: rifampin

INTERVENTIONS:
Drug: crizotinib — Treatment A: a single 250-mg dose of crizotinib will be administered in the fasted state on Day 1 as 1 × 50-mg and 2 × 100-mg Immediate Release Tablets.
Drug: rifampin — Treatment B: 600 mg once a day doses of rifampin will be orally administered after overnight fasting from Day 1 to Day 14.
Drug: crizotinib — Treatment B: A single 250-mg dose of crizotinib will be administered in the fasted state on Day 9 as 1 × 50-mg and 2 × 100-mg Immediate Release Tablets.

SUMMARY:
The purpose of this study is to estimate the effect of multiple doses of Rifampin on the single dose pharmacokinetics of Crizotinib in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non-child bearing potential subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Subjects with evidence of disease, conditions affecting drug absorption, treatment with other investigational drug within 30 days, history of regular alcohol consumption, and use of prescription , nonprescription drugs and dietary supplement within 7 days, and blood donation of 500 mL within 56 days.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, South Miami, Florida, United States

REFERENCES:
- [Derived] Xu H, O'Gorman M, Tan W, Brega N, Bello A. The effects of ketoconazole and rifampin on the single-dose pharmacokinetics of crizotinib in healthy subjects. Eur J Clin Pharmacol. 2015 Dec;71(12):1441-9. doi: 10.1007/s00228-015-1945-5. Epub 2015 Sep 18. PMID 26381275
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081016&StudyName=Estimation%20Of%20Effect%20Of%20Rifampin%20On%20Pharmacokinetics%20Of%20Crizotinib%20In%20Healthy%20Volunteers

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib 250 mg: Single oral dose of crizotinib 250 milligram (mg) immediate-release tablet (IRT) on Day 1 in first intervention period. A washout period of at least 14 days was maintained between each period.
- Crizotinib 250 mg + Rifampin 600 mg: Single oral dose of rifampin 600 mg tablet in fasted state from Day 1 to Day 14. A single oral dose of crizotinib 250 mg IRTs was administered on Day 9 in second intervention period. A washout period of at least 14 days was maintained between each period.
Period: First Intervention Period
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Started | 15 | 0
Completed | 14 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout Period (at Least 14 Days)
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Started | 14 | 0
Completed | 14 | 0
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Started | 0 | 14
Completed | 0 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive crizotinib 250 mg IRT first and then crizotinib 250 mg + rifampin 600 mg.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 38.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hours (hrs) post crizotinib dose in period 1 and Day 0, 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 2
Population: The pharmacokinetic (PK) parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Crizotinib 250 mg: Single oral dose of crizotinib 250 mg IRT in first intervention period [Treatment A (Reference)].
- Crizotinib 250 mg + Rifampin 600 mg: Single oral dose of rifampin 600 mg tablet in the fasted state from Day 1 to Day 14 and single oral dose of crizotinib 250 mg IRTs on Day 9 in second intervention period [Treatment B (Test)].
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 2192.00 (616.59) | 397.20 (106.12)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed AUC (0-∞) of crizotinib was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 18.21, 90% CI 2-sided [16.14 to 20.54]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 1 and Day 0, 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 2
Population: The PK parameter analysis population included all enrolled and treated participants who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng/mL | 102.10 (35.64) | 32.06 (11.23)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed Cmax of crizotinib was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 31.49, 90% CI 2-sided [26.43 to 37.51]

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 2103.00 (620.52) | 368.60 (101.93)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed AUClast of crizotinib was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 17.60, 90% CI 2-sided [15.48 to 20.02]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
hr | 5.0 [4.0 to 6.0] | 3.0 [2.0 to 5.0]

5. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
hr | 33.07 (6.96) | 48.23 (5.62)

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the body. Clearance obtained after oral dose CL/F is influenced by the fraction of the dose absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
L/hr | 118.80 (37.39) | 648.60 (164.95)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: L
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
L | 5940.0 (3242.9) | 45720.0 (15766.0)

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Crizotinib Metabolite (PF-06260182)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast) of crizotinib metabolite (PF-06260182).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 369.50 (119.58) | 20.28 (8.19)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed AUClast of PF-06260182 was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 5.49, 90% CI 2-sided [4.64 to 6.49]

9. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] for Crizotinib Metabolite (PF-06260182)
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞) of crizotinib metabolite (PF-06260182). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng*hr/mL | 378.60 (120.38) | 21.78 (8.98)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed AUC (0 - ∞) of PF-06260182 was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 5.75, 90% CI 2-sided [4.86 to 6.81]

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: as for outcome 2
Population: The PK parameter analysis population included all participants enrolled and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
hr | 5.0 [4.0 to 8.0] | 5.0 [2.0 to 6.0]

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
ng/mL | 29.88 (10.22) | 3.29 (1.23)
Statistical Analysis 1: Comparison: Crizotinib 250 mg vs Crizotinib 250 mg + Rifampin 600 mg; Natural log transformed Cmax of PF-06260182 was analyzed using a mixed effect model with treatment as a fixed effect and participant as a random effect. The adjusted mean differences and 90% CIs for the differences was exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 11.01, 90% CI 2-sided [9.02 to 13.45]

12. Secondary Outcome: Metabolite to Parent Ratio Area Under the Curve From Time Zero to Last Quantifiable Concentration (MRAUClast)
Description: Molar ratio of metabolite to parent area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (MRAUClast).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
Ratio | 0.1703 (0.0264) | 0.0533 (0.0112)

13. Secondary Outcome: Metabolite to Parent Ratio Area Under the Curve From Time Zero to Extrapolated Infinite Time [MRAUC (0 - ∞)]
Description: Molar ratio of metabolite to parent area under the curve from time zero to extrapolated infinite time [MRAUC (0-∞)].
Time Frame: 0 (pre-dose), 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 1 and Day 0, 0 (pre-dose) , 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72, 96 and 144 hrs post crizotinib dose in period 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
Ratio | 0.1676 (0.0271) | 0.0532 (0.0113)

14. Secondary Outcome: Metabolite to Parent Ratio Maximum Observed Plasma Concentration (MRCmax)
Description: Metabolite to parent molar ratio of maximum observed plasma concentration (MRCmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Number analyzed (Participants) | 15 | 14
Ratio | 0.2839 (0.0711) | 0.0996 (0.0382)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib 250 mg | Crizotinib 250 mg + Rifampin 600 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 250 mg (N=15) | Crizotinib 250 mg + Rifampin 600 mg (N=14)
Eye swelling (Eye disorders) | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.